CLINICAL TRIAL: NCT04820881
Title: Cerebrovascular Reactivity and Oxygen Metabolism as Markers of Neurodegeneration After Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Julie C. Chapman, Neuroscientist, Washington D.C. Veterans Affairs Medical Center
Other Study IDs: MIRB01897
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Measurement of cerebrovascular reactivity and oxygen metabolism before and after a single dose of 50mg sildenafil citrate. Diffusion tensor imaging, other structural imaging and cognitive testing will also be completed.
- Control Group: Measurement of cerebrovascular reactivity and oxygen metabolism before and after a single dose of 50mg sildenafil citrate. Diffusion tensor imaging, other structural imaging and cognitive testing will also be completed.

SUMMARY:
This grant award entitled, "Cerebrovascular Reactivity and Oxygen Metabolism as Markers for Neurodegeneration after Traumatic Brain Injury" (hereafter, "Neurovascular Study"), aims to determine if neurovascular contributors to neurodegeneration can serve as markers of the emergence or progression of degenerative processes after traumatic brain injury in middle-aged and older adults.

DETAILED DESCRIPTION:
This grant award entitled, "Cerebrovascular Reactivity and Oxygen Metabolism as Markers for Neurodegeneration after Traumatic Brain Injury" (hereafter, "Neurovascular Study"), aims to determine if neurovascular contributors to neurodegeneration can serve as markers of the emergence or progression of degenerative processes after traumatic brain injury in middle-aged and older adults. Primary outcomes are cerebrovascular reactivity (CVR), as measured by functional Magnetic Resonance Imaging (MRI) Blood Oxygen Level Dependent (BOLD) and cerebral metabolic rate of oxygen (CMRO2) as assessed by the novel MRI sequence called, "T-2 Relaxation-Under-Spin-Tagging" (TRUST). After the baseline primary endpoints are acquired, a single dose of sildenafil 50mg will be given to assess for the effects of a hypercapnia task on CVR and CMRO2. Other outcomes measured include additional imaging sequences (diffusion, ASL), volumetric analysis, and neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria (All Participants):

* Ages 50-80 years
* Eligible for Washington, DC Veterans Affairs Medical Center (VAMC) research participation
* Capacity to provide consent to participate in research (assessment made by study neurologist and PI)
* Ability to read and write English

Inclusion Criteria Case Group:

• History of traumatic brain injury of sufficient severity to have resulted in medical attention ascertained via the Ohio State University TBI Identification Questionnaire (OSU TBI-ID). TBI defined by Departments of Defense/Veterans Affairs (DoD/VA) criteria.

Inclusion Criteria Control Group:

• No history of traumatic brain injury of sufficient severity to have resulted in medical attention ascertained via the OSU TBI-ID, and no TBI based upon DOD/VA criteria.

Exclusion Criteria (All Participants):

* History of penetrating brain injury
* History or evidence of disabling neurological or psychiatric condition such as epilepsy (besides posttraumatic epilepsy), multiple sclerosis, hypoxic-ischemic encephalopathy, encephalitis, or schizophrenia
* History or evidence of cortical or subcortical stroke
* History or evidence of diabetes mellitus requiring therapy (Hemoglobin A1c > 9.0% for purposes of this study)
* History or evidence of uncontrolled hyperlipidemia. For the purposes of this study, "hyperlipidemia" will be defined as total cholesterol of 230 in the presence of either or both diabetes and hypertension and 300 in the absence of both of these conditions.

Statin therapy with normal cholesterol levels is allowed.

* History or evidence of uncontrolled hypertension (defined as systolic pressure > 160 and/or diastolic pressure > 110 mmHg), or hypotension (systolic pressure < 110 and/or diastolic pressure < 65 mmHg). Hypertension controlled with a single anti- hypertensive medication is allowed.
* Untreated atrial fibrillation
* Active tobacco use
* MRI incompatibility
* If a participant is currently or has previously taken a phosphodiesterase inhibitor (PDESi), then a two week washout period is required immediately prior to the evaluation visit.
* Use of nitrates

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle-aged and older adults with previous head injury experiencing current neurodegeneration.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular Reactivity (CVR) | Two years
  Cerebrovascular reactivity is the change in cerebral blood flow in response to a vasoactive stimulus, in this case hypercapnia induced by 5% carbon dioxide as measured by MRI BOLD
Cerebral Metabolic Rate of Oxygen (CMRO2) | Two years
  Cerebral metabolic rate of oxygen represents the amount of oxygen consumed as measured by the MRI T2-Relaxation-Under-Spin-Tagging (TRUST) sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Chapman, PsyD, Principal Investigator — Washington, DC VAMC
Locations (1):
- Washington, DC Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The grant that funds this study requires that de-identified data be submitted annually to the Federal Interagency Traumatic Brain Injury Research (FITBIR) Informatics System, of which the Department of Veterans Affairs is part. The FITBIR database, maintained by the National Institutes of Health, allows other researchers studying traumatic brain injury to apply for approval to utilize this previously collected, de-identified data for qualified research projects. Only de-identified data, which does not include anything that might directly identify participants, will be shared with FITBIR users who have been approved for research use.
Supporting Information: SAP, CSR
Time Frame: Time frame specified by the Federal Interagency Traumatic Brain Injury Research (FITBIR) Informatics Program.
Access Criteria: Access criteria specified by the Federal Interagency Traumatic Brain Injury Research (FITBIR) Informatics Program.
URL: http://fitbir.nih.gov